CLINICAL TRIAL: NCT02303769
Title: A Multicenter, Randomized, Double -Blind, Parallel, Comparative, Phase III Study to Investigate the Efficacy and Safety of GL2702 GLARS-NF1 Tablet in BPH Patients With LUTS
Brief Title: Study to Investigate the Efficacy and Safety of GL2702 GLARS-NF1tablet and Harnal-D - Tablet in BPH Patients With LUTS
Acronym: GL2702
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GL2702-301
Record Dates: First submitted 2014-11-11; First posted 2014-12-01 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Lower Urinary Track Syndrome; Harnal; Tamsulosin HCL 0.4mg
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tamsulosin HCL 0.2mg (Active Comparator): Harnal-D tablet (Tamsulosin HCL 0.2mg)
  Interventions: Drug: Tamsulosin HCL 0.2mg
- Tamsulosin HCL 0.4mg (Experimental): GL2702 GLARS-NF1 tablet (Tamsulosin HCL 0.4mg)
  Interventions: Drug: Tamsulosin HCL 0.4mg

INTERVENTIONS:
Drug: Tamsulosin HCL 0.4mg — Tamsulosin HCL 0.4mg once a day
  Other Names: GL2702 GLARS-NF1 Tablet
  Arms: Tamsulosin HCL 0.4mg
Drug: Tamsulosin HCL 0.2mg — Tamsulosin HCL 0.2mg once a day
  Other Names: Harmal D
  Arms: Tamsulosin HCL 0.2mg

SUMMARY:
Study to investigate the efficacy and safety of GL2702 GLARS-NF1tablet and Harnal-D - tablet in benign prostatic hyperplasia patients with lower urinary tract symptomatic

DETAILED DESCRIPTION:
GL2702 GLARS-NF1 tablet is controlled released formation which is made by GL Pharm Tech

ELIGIBILITY:
Inclusion Criteria:

* Over 50 years old, BPH diagnosted, Adult Male Subject
* IPSS ≥ 13 point
* PSA < 4ng/mL
* 5ml/sec < Qmax ≤ 15ml/sec

Exclusion Criteria:

* Prostatic cancer
* 250ml < PVR
* ALT or AST > 2 times (Upper Normal Range)
* Total Bilirubin > 1.5 times (Upper Normal Range)
* Treated with α-adrenalin receptor blocker within 2weeks before screening
* Treated with 5Alpha-Reductase Inhibitor within 6 months before screening
* Treated with phytotherapy within 2weeks before screening
* Treated with Anabolic Steroid within 6 months before screening

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in total International Prostate Symptom Score | 8 weeks

SECONDARY OUTCOMES:
Change from baseline to endpoint in total International Prostate Symptom Score | 4 weeks
Change from baseline to endpoint in voiding score | 4 weeks, 8 weeks
Change from baseline to endpoint in IPSS QoL | 4 weeks, 8 weeks
Change from baseline to endpoint in Qmax | 4 weeks, 8 weeks
Change from baseline to endpoint in PVR | 4 weeks, 8 weeks
Time to event/proportion of subjects with AUR | 8 weeks
Time to event/proportion of subjects undergoing BPH related prostatic surgery | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: You T Gun, MD, Principal Investigator — Eulji General Hospital
Locations (1):
- Eulji general hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No